CLINICAL TRIAL: NCT03046602
Title: Parental Real-life Experience During the Neonatal Transfer From Intensive Care Unit to Maternity Service of St Joseph Hospital
Brief Title: Parental Real-life Experience During the Neonatal Transfer
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: TransfereNN
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Neonatology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The transfer of newborn child from Intensive Care Unit to maternity is very stressfull for parents.This anxiety could have repercussion on parents adaptation on their new environment, on parent's role and also on their relaional interaction with the baby. As StJoseph hospital receives an important number of premature babies, the neonatology service aim to evaluate the real life experience of mothers during the transfer to set up improvement axes with hospital departments upstream.

ELIGIBILITY:
Inclusion Criteria:

* new born child transfered to St Joseph neonatology service
* Having stayed at least five days Intensive Care Unit
* Regardless of the term
* have to stay at least five days in neonatology

Exclusion Criteria:

* Non francophones parents
* Duration of predictable hospitalization of less than 5 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every new born child transfered to St Joseph neonatology service
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
mother's real life experience assessment during the transfer of new born child from intensive care unit to neonatology | day 3 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BEAUSSIER, Pharm-D, Study Director — CRC- GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No